CLINICAL TRIAL: NCT01886196
Title: Ibuprofen Supplementation After Resistance Training and Its Effects on Bone in Older Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Phil Chilibeck, Ph.D., University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12-256; DC0190GP (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2013-06-20; First posted 2013-06-25 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Sarcopenia; Osteoporosis
Keywords: elderly; women; exercise; pQCT; ibuprofen
MeSH Terms: conditions — Sarcopenia; Osteoporosis; Motor Activity | interventions — Anti-Inflammatory Agents, Non-Steroidal; Ibuprofen; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Non-steroidal anti-inflammatory drug (Experimental): ibuprofen after exercise training sessions (400 mg, 3 times per week for 9 months)
  Interventions: Drug: Non-steroidal anti-inflammatory drug (Ibuprofen); Behavioral: Resistance exercise
- placebo (Placebo Comparator): placebo after exercise training sessions(3 times per week for 9 months)
  Interventions: Other: placebo; Behavioral: Resistance exercise
- resistance exercise (Experimental): 3 sets of 8-12 repetitions of resistance exercises focused on distal radius to be performed 3 times/week for 9 months
  Interventions: Drug: Non-steroidal anti-inflammatory drug (Ibuprofen); Other: placebo
- flexibility training (Sham Comparator): flexibility training to be performed 3 days/week for 1 hour for 9 months
  Interventions: Other: placebo; Behavioral: Flexibility training

INTERVENTIONS:
Drug: Non-steroidal anti-inflammatory drug (Ibuprofen) — 400mg of ibuprofen administered after exercise training session 3 days per week
  Other Names: Ibuprofen
  Arms: Non-steroidal anti-inflammatory drug; resistance exercise
Other: placebo — placebo designed to mimic experimental drug (ibuprofen)
  Arms: flexibility training; placebo; resistance exercise
Behavioral: Resistance exercise — 3 sets of 8-12 repetitions of resistance exercise (full body with a focus on the distal radius) completed 3 days/week under supervision in the research gym
  Arms: Non-steroidal anti-inflammatory drug; placebo
Behavioral: Flexibility training — 3 days of full body stretching program (approximately 1 hour) to be performed at participants home unsupervised
  Arms: flexibility training

SUMMARY:
Inflammation increases with aging and is implicated in the reduction of bone mass, muscle mass, and strength. Resistance training is safe and effective for increasing muscle mass and strength in older adults,however resistance training by itself cannot suppress inflammation. Ibuprofen is a non-steroidal anti-inflammatory drug that may provide benefits to muscle mass and strength when given after resistance training sessions in older adults; however, more evidence is required to confirm effects across the lifespan. The objectives are to determine the effect of 9 months of exercise training and ibuprofen supplementation, compared to placebo, in older women (≥65years)on the following dependent variables:

* bone density, geometry, and architecture
* muscle mass and strength
* balance

DETAILED DESCRIPTION:
The aim of our study is to create new evidence about the effectiveness and safety of non-steroid anti-inflammatory supplementation (i.e. ibuprofen) combined with exercise to influence positively bone and muscle health in women aged 65 years and older. With aging, there is a significant decrease in bone mineral, muscle mass, and strength, which increases the risk of falls, injuries and fracture especially for women. Direct and indirect health costs associated with osteoporosis and sarcopenia (defined as "muscle wasting") are in the billions of dollars and escalating as the proportion of older adults in Canada grows. Low-grade inflammation is a main contributing factor to bone and muscle deterioration with aging but is mitigated by anti-inflammatory drug use. Recent evidence shows resistance exercise training combined with a non-steroidal anti-inflammatory drug (ibuprofen) is effective for increasing bone mineral density in young women. No study has addressed directly the effects of ibuprofen use following resistance exercise on bone and muscle in older women, the population at greatest risk of developing osteoporosis. The primary purpose of this study is to investigate the safety and multiple effects of ibuprofen ingestion following supervised resistance exercise training on bone and muscle in older women (≥65y).

PRIMARY HYPOTHESES: Ibuprofen combined with resistance training will maintain hip and lumbar spine areal bone mineral density in older women. Secondary hypotheses are that bone structural properties in the hip and wrist, and muscle mass and strength will be improved by supplementing ibuprofen after resistance training sessions.

RESEARCH PLAN: The study will use a repeated measures, parallel group randomized design where 100 women (≥65 y) will be randomized to one of 4 groups: 1) Exercise and ibuprofen (400 mg immediately after exercise); 2) Exercise and ibuprofen placebo; 3) Placebo exercise and ibuprofen, 4) Placebo exercise and ibuprofen placebo. Women will participate in the exercise sessions 3 days per week. The intervention will be 9 months in duration. Dual energy X-ray absorptiometry (DXA) will be used to assess hip and lumbar spine areal bone mineral density, as well as geometric changes in hip structure, and whole body lean tissue (i.e. muscle) mass. Peripheral quantitative computed tomography (pQCT) and high-resolution-pQCT will allow us to investigate detailed changes in bone microarchitecture at the wrist and muscle cross-sectional area in the forearm in response to the intervention. Safety will be addressed by closely monitoring adverse events.

RELEVANCE: This pilot study potentially drives a novel post-market use of ibuprofen. In addition, it permits our developing research team a foray into preliminary data collection to inform a larger randomized controlled trial (RCT) application to CIHR.

ELIGIBILITY:
Inclusion Criteria:

* women >65yrs

Exclusion Criteria:

* high risk of fracture
* use of bisphosphonates, hormone replacement therapy, selective estrogen receptor modulators, PTH, or calcitonin within the past 12 months
* taking medications that affect bone mineral metabolism
* have diseases that are known to affect bone mineral metabolism
* have severe osteoarthritis
* currently a smoker
* currently participating in moderate-vigorous resistance-exercise training more than once per week

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
change from baseline in aBMD of the proximal femur and lumbar spine at 9 months | baseline and 9 months
  areal bone mineral density of the proximal femure and lumbar spine assessed by dual energy x-ray absorptiometry

SECONDARY OUTCOMES:
change from baseline in femoral neck section modulus at 9 months | baseline and 9 months
  femoral neck section modulus assessed by dual energy x-ray absorptiometry
change from baseline in distal radius Bone Strength Index at 9 months | baseline and 9 months
  distal radius Bone Strength Index assessed by high resolution peripheral quantitative computed tomography
change from baseline in radial shaft Stress Strain Index at 9 months | baseline and 9 months
  radial shaft Stress Strain Index assessed by peripheral quantitative computed tomography
change from baseline in radial shaft muscle cross-sectional area at 9 months | baseline and 9 months
  radial shaft muscle cross-sectional area assessed by peripheral quantitative computed tomography
change from baseline in total body lean tissue mass at 9 months | baseline and 9 months
  total body lean tissue mass assessed by dual energy x-ray absorptiometry
change from baseline in muscular strength at 9 months | baseline and 9 months
  muscular strength assessed by 1 repetition maximum bicep curl and leg press
change from baseline in balance performance at 9 months | baseline and 9 months
  balance performance assessed by tandem walk on balance board

OTHER OUTCOMES:
number of participants with adverse events as a measure of safety and number of participants wit adverse events as a measure of safety and tolerability | continuously throughout 9 months
  adverse events as reported by participants and charted on 'adverse events' form

CONTACTS AND LOCATIONS:
Overall Officials: Philip D Chilibeck, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- College of Kinesiology, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krentz JR, Quest B, Farthing JP, Quest DW, Chilibeck PD. The effects of ibuprofen on muscle hypertrophy, strength, and soreness during resistance training. Appl Physiol Nutr Metab. 2008 Jun;33(3):470-5. doi: 10.1139/H08-019. PMID 18461099